CLINICAL TRIAL: NCT05888324
Title: Factors Associated With the Onset of Chronic Headaches in Patients Who Received a Blood Patch, Following an Accidental Dural Puncture During Post Partum Period
Brief Title: Factors Associated With the Onset of Chronic Headaches in Patients Who Received a Blood Patch in Post Partum
Acronym: CHROBLOOD
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220572; 022-A00933-40 (Other: France : ANSM)
Record Dates: First submitted 2022-11-14; First posted 2023-06-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Blood Patch; Post-Dural Puncture Headache
Keywords: Post Dural puncture headache; Epidural blood patch; Chronic headache; Epidural analgesia; Obstetric anaesthesia
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with PDPH after epidural analgesia for labor, requiring BP: Patients with PDPH after epidural analgesia for labor, requiring BP
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires by phone at 1 and 6 months after inclusion

SUMMARY:
The purpose of this study is to identify possible links between conditions for carrying out a blood patch (BP) to treat accidental post dural puncture acute headache (PDPH) in the early post partum period and occurrence of chronic headaches at 1 and 6 months.

DETAILED DESCRIPTION:
It is established that accidental dural puncture promotes the onset of chronic headaches in 25 to 60% of cases but the risk factors for the occurrence of this event are not known.

To identify those risk factors, the investigators will analyze the initial conditions of the accidental breach, the initial manifestations of the PDPH, the methods of carrying out the BP and the patient data.

In this study, the investigators will evaluate (phone questionnaire and score) incidence of chronic headaches at 1 month and 6 months after the realization of a blood patch, incidence of chronic low back pain, impact on daily life, incidence of late recurrences of PDPH, incidence of early and distant complications

In case of failure of effectiveness of the first blood patch, the investigators will search for associated factors: patient data, mode of delivery, initial PDPH, conditions for carrying out the BP.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old,
* Vaginal delivery or caesarean section with epidural at the Port Royal maternity ward,
* Collection of non-opposition after oral and written information,

Exclusion Criteria:

* Patient under curatorship or guardianship
* Not speaking/understanding French
* BP performed in another indication
* Benefiting from the AME (state medical aid)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vaginal delivery or caesarean section with epidural at the Port Royal maternity ward
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Description of the conditions of the accidental breach | Immediately after BloodPatch procedure
  Data collection of diagnosis of the accidental breach :
  * noted with the needle,
  * intrathecal passage,
  * postpartum positional headaches,
  * intrathecal catheter
Time to onset | Immediately after BloodPatch procedure
  Description of the initial manifestations of post dural puncture acute headache (PDPH) : nature of PDPH
Positional | Immediately after BloodPatch procedure
  Description of the initial manifestations of post dural puncture acute headache (PDPH) : nature of PDPH
Neck pain | Immediately after BloodPatch procedure
  Description of the initial manifestations of post dural puncture acute headache (PDPH) : nature of PDPH
Analog visual scale (AVS) | Immediately after BloodPatch procedure
  Description of the initial manifestations of post dural puncture acute headache (PDPH) : nature of PDPH
Neurosensory disorders | Immediately after BloodPatch procedure
  Description of the initial manifestations of post dural puncture acute headache (PDPH) : nature of PDPH
Completion time after childbirth | Immediately after BloodPatch procedure
  Description of the methods of carrying out the BloodPatch (BP)
Volume injected | Immediately after BloodPatch procedure
  Description of the methods of carrying out the BloodPatch (BP)
Height of puncture compared to the initial breach | Immediately after BloodPatch procedure
  Description of the methods of carrying out the BloodPatch (BP)
Paresthesias | Immediately after BloodPatch procedure
  Description of the methods of carrying out the BloodPatch (BP)
Adverse events | Immediately after BloodPatch procedure
  Description of the methods of carrying out the BloodPatch (BP)
Duration of strict decubitus in the immediate afterglow | Immediately after BloodPatch procedure
  Description of the methods of carrying out the BloodPatch (BP)
Age | Immediately after BloodPatch procedure
  Patient data collection
Height | Immediately after BloodPatch procedure
  Patient data collection
Weight | Immediately after BloodPatch procedure
  Patient data collection
Parity | Immediately after BloodPatch procedure
  Patient data collection
Mode of delivery | Immediately after BloodPatch procedure
  Patient data collection
History of headaches or migraines before pregnancy | Immediately after BloodPatch procedure
  Patient data collection
Initial treatment (before 1st BP) | Immediately after BloodPatch procedure
  Patient data collection NSAIDs and analgesics, sphenopalatine ganglion block, ACTH, caffeine, other
Imaging | 1 month after last BloodPatch procedure
  Patient data collection
Lumbar punction | 1 month after last BloodPatch procedure
  Patient data collection
Other examinations if performed | 1 month after last BloodPatch procedure
  Patient data collection
Complications during the initial postpartum stay | Immediately after BloodPatch procedure
  Patient data collection
Analog visual scale (AVS) | Immediately after BloodPatch procedure
  Patient data collection - Initial efficacy
Analog visual scale (AVS) | 1 day after BloodPatch procedure
  Patient data collection - Initial efficacy
Analog visual scale (AVS) | At exit of the hospital, up to 2 weeks
  Patient data collection - Initial efficacy

SECONDARY OUTCOMES:
Number of patients with chronic headaches | Month 1
  Score - phone questionnaire
Number of patients with chronic headaches | Month 6
  Score - phone questionnaire
Number of patients with chronic low back pain | Month 1
  Score - phone questionnaire
Number of patients with chronic low back pain | Month 6
  Score - phone questionnaire
Modified Headache Impact Questionnaire (HIT) | Month 1
  Impact on daily life - Phone questionnaire - Headaches : "Yes/No" Low back pain, "never/rarely/from time to time/often/all the time"
Modified Headache Impact Questionnaire (HIT) | Month 6
  Impact on daily life - Phone questionnaire - Headaches : "Yes/No" Low back pain, "never/rarely/from time to time/often/all the time"
Number of patients with late recurrence of typical post dural puncture acute headache (PDPH) | Month 1
  Score - phone questionnaire
Number of patients with late recurrence of typical post dural puncture acute headache (PDPH) | Month 6
  Score - phone questionnaire
Number of patients who have been rehospitalized | Month 1
  Score - phone questionnaire
Number of patients who have been rehospitalized | Month 6
  Score - phone questionnaire
Number of patients consulted for headaches | Month 1
  Score - phone questionnaire
Number of patients consulted for headaches | Month 6
  Score - phone questionnaire
Number of patients who received complementary treatments | Month 1
  Score - phone questionnaire
Number of patients who received complementary treatments | Month 6
  Score - phone questionnaire
Patient data collection | Month 1
  In case of failure of efficacy of the 1st BP: patient data, mode of delivery, initial Post dural puncture acute headache (PDPH), conditions for carrying out the BP
Patient data collection | Month 6
  In case of failure of efficacy of the 1st BP: patient data, mode of delivery, initial Post dural puncture acute headache (PDPH), conditions for carrying out the BP

CONTACTS AND LOCATIONS:
Overall Officials: Catherine FISCHER, MD, Principal Investigator — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Port-Royal Maternity ward - Cochin Hopsital - APHP, Paris, Île-de-France Region, France